CLINICAL TRIAL: NCT01701427
Title: Hyperalgesia After Deep Electrical Stimulation in Pain Free Subjects
Brief Title: Pain After Deep Electrical Stimulation in the Groin in Pain Free Subjects
Acronym: HADES-1
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, M.D., Rigshospitalet, Denmark
Other Study IDs: H-1-2012-035
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Persistent Postherniotomy Pain
Keywords: Hyperalgesia; Persistent pain; deep pain; electrical stimulation; groin hernia
MeSH Terms: conditions — Hyperalgesia; Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: 1. Healthy, un-operated, groin-hernia free, pain-free and medicinal free males

SUMMARY:
Sensory disturbances in persistent postherniotomy pain, include hyperalgesia from deeper structures as well as the skin. Whether this is one combined pain syndrome, where for instance deep pain leads to cutaneous hyperalgesia, or two isolated synchronous pain conditions, is unknown. By Giving pain free subjects an intense non-harmful electrical stimulation in deeper tissues in the groin and recording the skin sensory function, this hypothesis will be tested

ELIGIBILITY:
Inclusion Criteria:

* male, age >18 yr, pain-free, caucasian

Exclusion Criteria:

* previous groin surgery, groin hernia, sensory disturbaces, use of painmedication, drug or alcohol abuse.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy young men.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in skin pain detection threshold before and during deep electrical pain stimulation. | 14 days
  Heat pain detection threshold by use of a Thermotester (Somedic AS Sweden) is assessed before and during deep electrical pain stimulation (6 of 10 point on a NRS scale. Deep pain stimulation is performed by two needle electrodes, placed under ultrasound guidance, 5 mm apart in various tissue and locations in the groin:
  1. Musculus rectus abdominis dxt. ( 10 cm craniel to the external inguinal ring) - Subcutaneous, and muscular stimulation.
  2. Spina iliaca anterior superior dxt. ( 2 cm lateral to the ilica spine) - subcutaneous, m obliquus externus and nervns ilioinguinalis stimulation.
  3. External inguinal ring - subcutaneous and funicle stimulation.

SECONDARY OUTCOMES:
Test-retest of primary outcome | 14 days
  The primay and additional assesments are re-measured 14 days after the primary assemssment to allow evaluation of test-retest reliability.

OTHER OUTCOMES:
deep electrical and pain detection thresholds | 14 days
  The detection- and pain detection thresholds to electrical stimulation will be assessed. An up-n-down staircase stimulation of single oulses of 0.04 mSeconds with increasing mA from 0.1 to a maximum of 60 mA is used. A total of 10 thresholds is recorded in the following locations.
  Musculus rectus abdominis dxt. ( 10 cm craniel to the external inguinal ring) - Subcutaneous, and muscular stimulation.
  Spina iliaca anterior superior dxt. ( 2 cm lateral to the ilica spine) - subcutaneous, m obliquus externus and nervns ilioinguinalis stimulation.
  External inguinal ring - subcutaneous and funicle stimulation. Musculus rectus abdominis sin. ( 10 cm craniel to the external inguinal ring) - Subcutaneous, and muscular stimulation.
warmth and mechanical detection and pain detection thresholds | 14 days
  warmth and mechanical detection and pain detection thresholds are recorded in the right and left groin and right lower arm. A total of 10 repated mesures for each parameter is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Section for Surgical Pathophysiology, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Aasvang EK, Werner MU, Kehlet H. Referred pain and cutaneous responses from deep tissue electrical pain stimulation in the groin. Br J Anaesth. 2015 Aug;115(2):294-301. doi: 10.1093/bja/aev170. Epub 2015 Jun 12. PMID 26071091